CLINICAL TRIAL: NCT02000843
Title: Tympanoplasty -- Conchal Cavum Approach
Brief Title: Tympanoplasty Using Conchal Cavum Approach and Conchal Pericondrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H13-03261
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Perforation of Eardrum.
Keywords: perforation; tympanoplasty; conchal cavum approach; perichondrium/ cartilage; scar
MeSH Terms: conditions — Tympanic Membrane Perforation; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- perichondrium graft perforation (Other): tympanoplasty -- conchal cavum approach is used.
  Interventions: Procedure: tympanoplasty -- conchal cavum approach

INTERVENTIONS:
Procedure: tympanoplasty -- conchal cavum approach — Incision is made inside the ear canal. It is extended into the conchal cavum. The incision allows a direct approach to the eardrum, and also allow easy harvesting of the perichondrium to be used as graft material.

SUMMARY:
Tympanoplasty -- conchal cavum approach is a modification of Heermann endural approach to repair broken eardrums. The Heermann approach is a well recognized procedure, in common clinical practise for years.

The new approach has been used in patients after informed consent was obtained from each patient.

DETAILED DESCRIPTION:
From 2010 to 2013, a total of 96 patients had the procedure. The data are entered, and analyzed. All identifiable information would be hidden.

This application is to obtain patients' consent for release and publication of the data. Patients would be assured their identities are protected.

ELIGIBILITY:
Inclusion Criteria:

* All patients with informed consent

Exclusion Criteria:

* Patients without consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
success rate of repair of eardrum | one year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Man, MD FRCS(C), Principal Investigator — UBC
Locations (1):
- Christopher Man, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Mohamad SH, Khan I, Hussain SS. Is cartilage tympanoplasty more effective than fascia tympanoplasty? A systematic review. Otol Neurotol. 2012 Jul;33(5):699-705. doi: 10.1097/MAO.0b013e318254fbc2. PMID 22643445
- [Derived] Man SC, Nunez DA. Tympanoplasty--conchal cavum approach. J Otolaryngol Head Neck Surg. 2016 Jan 6;45:1. doi: 10.1186/s40463-015-0113-3. PMID 26739478